CLINICAL TRIAL: NCT02875834
Title: A Phase 3 Multicenter, Prospective, Randomized, Double-blind, Placebo-controlled Study to Investigate the Safety and Efficacy of ZS, in Patients With Hyperkalemia-HARMONIZE Global
Brief Title: A Study to Investigate the Safety and Efficacy of ZS in Patients With Hyperkalemia
Acronym: HARMONIZE GL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D9480C00002
Record Dates: First submitted 2016-07-22; First posted 2016-08-23 (Estimated); Results first posted 2020-08-19 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Hyperkalemia
MeSH Terms: conditions — Hyperkalemia | interventions — sodium zirconium cyclosilicate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sodium Zirconium Cyclosilicate (ZS) 5g (Experimental): Suspension administered 5g orally once daily for 28 days after the first 48-hour open label initial phase.
  Interventions: Drug: Sodium Zirconium Cyclosilicate (ZS) 5g
- Sodium Zirconium Cyclosilicate (ZS) 10g (Experimental): Suspension administered 10g orally once daily for 28 days after the first 48-hour open label initial phase.
  Interventions: Drug: Sodium Zirconium Cyclosilicate (ZS) 10g
- Placebo (Placebo Comparator): Suspension administered orally placebo once daily for 28 days after the first 48-hour open label initial phase.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sodium Zirconium Cyclosilicate (ZS) 10g — Suspension administered 10g orally three times per day, in the first 48-hour of the study for all patients (48-hour open label initial phase)
  Arms: Sodium Zirconium Cyclosilicate (ZS) 10g
Drug: Sodium Zirconium Cyclosilicate (ZS) 5g — Suspension administered 5g orally once daily for 28 days after the first 48-hour open label initial phase.
  Arms: Sodium Zirconium Cyclosilicate (ZS) 5g
Drug: Sodium Zirconium Cyclosilicate (ZS) 10g — Suspension administered 10g orally once daily for 28 days after the first 48-hour open label initial phase.
  Arms: Sodium Zirconium Cyclosilicate (ZS) 10g
Drug: Placebo — Suspension administered orally placebo once daily for 28 days after the first 48-hour open label initial phase.
  Arms: Placebo

SUMMARY:
To evaluate the efficacy of two different doses (5 and 10 g) of ZS orally administered once daily (qd) vs placebo in maintaining normokalemia in initially hyperkalemic patients having achieved normokalemia following two days of initial ZS therapy (10g TID).

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures
* Female and male patients aged ≥18 and ≤ 90 years
* Two consecutive i-STAT potassium values, measured 60-minutes (± 10 minutes) apart, both ≥ 5.1 mmol/l and measured within 1 day of the first ZS dose on 48-hour open-label initial phase Day 1
* Ability to have repeated blood draws or effective venous catheterization
* Female patients must be 1 year post-menopausal, surgically sterile, or using an acceptable method of contraception for the duration of the study and for 3 months after the last dose of ZS/matching placebo to prevent pregnancy.

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study
* Participation in another clinical study with an investigational product during the last 3 months
* Pseudohyperkalemia signs and symptoms
* Patients treated with lactulose, xifaxan (rifaximin) or other non-absorbed antibiotics for hyperammonemia within 7 days prior to the first dose of study drug
* Patients treated with resins,calcium acetate,calcium carbonate, or lanthanum carbonate,within 7 days prior to the first dose of study drug
* Patients with a life expectancy of less than 3 months
* Patients who are severely physically or mentally incapacitated and who in the opinion of investigator are unable to perform the subjects' tasks associated with the protocol
* Female patients who are pregnant, lactating, or planning to become pregnant
* Patients with diabetic ketoacidosis
* Presence of any condition which, in the opinion of the investigator, places the patient at undue risk or potentially jeopardizes the quality of the data to be generated
* Known hypersensitivity or previous anaphylaxis to ZS or to components thereof
* Patients with cardiac arrhythmias that require immediate treatment
* Patients on dialysis
* Patients who are blood donors should not donate blood during the study and for 3 months following their last dose of ZS

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2018-02-14 (Actual); Study Completion 2018-02-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (34):
- Japan (13):
  - Research Site, Chiba
  - Research Site, Hanyu-shi
  - Research Site, Hitachi-Naka
  - Research Site, Ina-shi
  - Research Site, Kanazawa
  - Research Site, Koga-shi
  - Research Site, Matsudo-shi
  - Research Site, Nagoya
  - Research Site, Shimajiri-gun
  - Research Site, Shizuoka
  - Research Site, Toride-shi
  - Research Site, Toyohashi
  - Research Site, Yakushi
- Russia (5):
  - Research Site, Krasnoyarsk
  - Research Site, Moscow
  - Research Site, Saint Petersburg
  - Research Site, Yaroslavl
  - Research Site, Yekaterinburg
- South Korea (12):
  - Research Site, Anyang-si
  - Research Site, Bucheon-si
  - Research Site, Busan
  - Research Site, Cheongju-si
  - Research Site, Goyang-si
  - Research Site, Gwangju
  - Research Site, Hwaseong-si
  - Research Site, Incheon
  - Research Site, Seoul
  - Research Site, Suwon
  - Research Site, Uijeongbu-si
  - Research Site, Wŏnju
- Taiwan (4):
  - Research Site, Hualien City
  - Research Site, New Taipei City
  - Research Site, Taichung
  - Research Site, Taipei

REFERENCES:
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4401&filename=d9480c00002-sap-ed-2_Redacted_CTT.PDF
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4401&filename=d9480c00002-csp-v3_Redacted_CTT.PDF

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 42 centers within Japan, Russia, South Korea, and Taiwan.
Pre-assignment Details: the study consisted of two phases: an open-label phase (single arm, 48 hours, ZS 10 g TID; OLP) and a randomized treatment phase (3 arms, 28 days; RTP). 267 patients entered OLP. Out of these, 248 endered RTP and were randomized to placebo, ZS 5 g QD or ZS 10 g QD in a 1:2:2 ratio.
Groups:
- Sodium Zirconium Cyclosilicate (ZS) 10g Tid: Suspension administered 10g orally 3 times per day for the first 48-hour open label initial phase.
Period: Open-label Phase
Arm/Group | Sodium Zirconium Cyclosilicate (ZS) 10g Tid | Sodium Zirconium Cyclosilicate (ZS) 5g | Sodium Zirconium Cyclosilicate (ZS) 10g | Placebo
Started | 267 | 0 | 0 | 0
Completed | 260 | 0 | 0 | 0
Not Completed | 7 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 0 | 0
Not completed — (Not collected) | 4 | 0 | 0 | 0
Period: Randomized Treatment Phase
Arm/Group | Sodium Zirconium Cyclosilicate (ZS) 10g Tid | Sodium Zirconium Cyclosilicate (ZS) 5g | Sodium Zirconium Cyclosilicate (ZS) 10g | Placebo
Started | 0 (No subjects were randomized in 10g TID group in RTP.) | 99 (99 subjects were randomized in 5g QD group in RTP.) | 99 (99 subjects were randomized in 10g QD group in RTP.) | 50 (50 subjects were randomized in placebo group in RTP.)
Completed | 0 | 85 | 88 | 41
Not Completed | 0 | 14 | 11 | 9
Not completed — Withdrawal by Subject | 0 | 3 | 1 | 0
Not completed — Protocol Violation | 0 | 2 | 0 | 0
Not completed — (Not collected) | 0 | 9 | 10 | 9

BASELINE CHARACTERISTICS:
Population: In RTP there were no subjects analyzed in Sodium Zirconium Cyclosilicate (ZS) 10g tid arm. In OLP, only ZS 10 g TID arm was present. All subjects in RTP took part in OLP.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sodium Zirconium Cyclosilicate (ZS) 10g Tid | Sodium Zirconium Cyclosilicate (ZS) 5g | Sodium Zirconium Cyclosilicate (ZS) 10g | Placebo | Total
Number analyzed (Participants) | 267 | 99 | 99 | 50 | 515
Age, Continuous [Mean (Standard Deviation); unit: Years] — All subjects in RTP took part in OLP. Thus, the Totals are calculated using replicated measurements. Population: RTP: For the 28-day randomized treatment study phase, the Full Analysis Set (FAS) will include all patients who are randomized to the 28-day randomized treatment study phase.
  Years | 67.8 (10.80) | 66.7 (11.40) | 68.0 (10.18) | 69.4 (10.26) | 67.7 (10.70)
Sex: Female, Male [Count of Participants; unit: Participants] — All subjects in RTP took part in OLP. Thus, the Totals are calculated using replicated measurements.
  Participants
    Female | 96 | 36 | 38 | 14 | 184
    Male | 171 | 63 | 61 | 36 | 331
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — All subjects in RTP took part in OLP. Thus, the Totals are calculated using replicated measurements.
  Participants
    Hispanic or Latino | 2 | 0 | 1 | 1 | 4
    Not Hispanic or Latino | 265 | 99 | 98 | 49 | 511
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — All subjects in RTP took part in OLP. Thus, the Totals are calculated using replicated measurements.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
    Asian | 227 | 87 | 86 | 43 | 443
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 0 | 0
    White | 40 | 12 | 13 | 7 | 72
    More than one race | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Country [Count of Participants; unit: Participants] — All subjects in RTP took part in OLP. Thus, the Totals are calculated using replicated measurements.
  Participants
    Japan | 68 | 26 | 27 | 13 | 134
    Korea | 121 | 46 | 45 | 23 | 235
    Russia | 40 | 12 | 13 | 7 | 72
    Taiwan | 38 | 15 | 14 | 7 | 74

OUTCOME MEASURES:

1. Primary Outcome: Least Square Mean S-K Level on Days 8-29
Description: Comparison between placebo and the active ZS treatment groups (each dose group will be sequentially compared with placebo, starting with the highest and ending with the lowest dose) with regard to the mean S-K level during the 28-day randomized treatment study phase Days 8-29. The results in the table below are presented for RTP.
Time Frame: Through 28-day randomized treatment study phase day 8-29.
Population: Full Analysis Set
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Sodium Zirconium Cyclosilicate (ZS) 10g Tid | Sodium Zirconium Cyclosilicate (ZS) 5g | Sodium Zirconium Cyclosilicate (ZS) 10g | Placebo
Number analyzed (Participants) | 0 | 99 | 99 | 50
mmol/L |  | 4.811 [4.685 to 4.940] | 4.381 [4.265 to 4.501] | 5.321 [5.155 to 5.493]
Statistical Analysis 1: Comparison: Sodium Zirconium Cyclosilicate (ZS) 5g vs Placebo; Results derived from a mixed effects model of log-transformed S-K levels. Fixed effects are: treatment group; visit; treatment-by-visit interaction; baseline S-K values (OLP and RTP); baseline eGFR; age category; country; baseline RAAS inhibitor, chronic kidney disease, heart failure, and diabetes mellitus statuses. Patient is a random effect. p-values given are for differences of LSMEANS. The back-transformation is to the original scale of the S-K measurement; Test type: Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.904, 95% CI 2-sided [0.876 to 0.933]
Statistical Analysis 2: Comparison: Sodium Zirconium Cyclosilicate (ZS) 10g vs Placebo; Test type: Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.823, 95% CI 2-sided [0.797 to 0.850]

2. Secondary Outcome: Proportion of Patients Achieving Normokalemia
Description: Proportion of patients who achieve normokalemia during the initial phase at 24 and 48 hours. The results in the table below are presented for OLP. (h=hours).
Time Frame: Through 48-hour initial phase.
Population: Full Analysis Set
Measure: Number; unit: Participants
Arm/Group | Sodium Zirconium Cyclosilicate (ZS) 10g Tid | Sodium Zirconium Cyclosilicate (ZS) 5g | Sodium Zirconium Cyclosilicate (ZS) 10g | Placebo
Number analyzed (Participants) | 267 | 0 | 0 | 0
Participants
  Normokalemic at 24h | 169 |  |  |
  Not Normokalemic at 24h | 93 |  |  |
  Missing at 24h | 5 |  |  |
  Normokalemic at 48h | 238 |  |  |
  Not Normokalemic at 48h | 22 |  |  |
  Missing at 48h | 7 |  |  |

3. Secondary Outcome: Exponential Rate of Change in S-K Levels
Description: Exponential rate of change in S-K levels (blood) during the 48-hour open-label initial phase. The results in the table below are presented for OLP.
Time Frame: Through 48-hour initial phase.
Population: Full Analysis Set
Measure: Mean (Standard Error); unit: log(mmol/L)/h
Arm/Group | Sodium Zirconium Cyclosilicate (ZS) 10g Tid | Sodium Zirconium Cyclosilicate (ZS) 5g | Sodium Zirconium Cyclosilicate (ZS) 10g | Placebo
Number analyzed (Participants) | 267 | 0 | 0 | 0
log(mmol/L)/h | -0.004 (0.0001) |  |  |

4. Secondary Outcome: Absolute Change From Baseline in S-K Levels
Description: Absolute change from baseline in S-K levels at all measured time intervals. The results in the table below are presented for OLP.
Time Frame: Through 48-hour initial phase.
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Sodium Zirconium Cyclosilicate (ZS) 10g Tid | Sodium Zirconium Cyclosilicate (ZS) 5g | Sodium Zirconium Cyclosilicate (ZS) 10g | Placebo
Number analyzed (Participants) | 267 | 0 | 0 | 0
mmol/L
  OLP Day 1-1h post-first dose absolute change | -0.19 (0.444) |  |  |
  OLP Day 1-2h post-first dose absolute change | -0.48 (0.452) |  |  |
  OLP Day 1-4h post-first dose absolute change | -0.57 (0.494) |  |  |
  OLP Day 2-24h absolute change: number analyzed (Participants) | 262 | 0 | 0 | 0
  OLP Day 2-24h absolute change | -0.81 (0.398) |  |  |
  OLP Day 2-1h post-first dose absolute change: number analyzed (Participants) | 261 | 0 | 0 | 0
  OLP Day 2-1h post-first dose absolute change | -0.91 (0.445) |  |  |
  OLP Day 3-48h absolute change: number analyzed (Participants) | 260 | 0 | 0 | 0
  OLP Day 3-48h absolute change | -1.28 (0.499) |  |  |

5. Secondary Outcome: Percentage Change From Baseline in S-K Levels
Description: Percentage change from baseline in S-K levels at all measured time intervals. The results in the table below are presented for OLP.
Time Frame: Through 48-hour initial phase.
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Sodium Zirconium Cyclosilicate (ZS) 10g Tid | Sodium Zirconium Cyclosilicate (ZS) 5g | Sodium Zirconium Cyclosilicate (ZS) 10g | Placebo
Number analyzed (Participants) | 267 | 0 | 0 | 0
Percentage change
  OLP Day 1-1h post-first dose percentage change | -3.26 (7.949) |  |  |
  OLP Day 1-2h post-first dose percentage change | -8.29 (7.792) |  |  |
  OLP Day 1-4h post-first dose percentage change | -9.88 (8.494) |  |  |
  OLP Day 2-24h percentage change: number analyzed (Participants) | 262 | 0 | 0 | 0
  OLP Day 2-24h percentage change | -14.08 (6.479) |  |  |
  OLP Day 2-1h post-first dose percentage change: number analyzed (Participants) | 261 | 0 | 0 | 0
  OLP Day 2-1h post-first dose percentage change | -15.84 (7.243) |  |  |
  OLP Day 3-48h percentage change: number analyzed (Participants) | 260 | 0 | 0 | 0
  OLP Day 3-48h percentage change | -22.16 (7.812) |  |  |

6. Secondary Outcome: Proportion of Patients Remaining Normokalemic
Description: The proportion of patients who remain normokalemic (as defined by S-K between 3.5-5.0 mmol/l, inclusive) at the end of the 28-day randomized treatment study phase and during the 28-day randomized treatment study phase. The results in the table below are presented for RTP.
Time Frame: Through 28-day randomized treatment study phase day 8-29.
Population: Full Analysis Set
Measure: Number; unit: Participants
Arm/Group | Sodium Zirconium Cyclosilicate (ZS) 10g Tid | Sodium Zirconium Cyclosilicate (ZS) 5g | Sodium Zirconium Cyclosilicate (ZS) 10g | Placebo
Number analyzed (Participants) | 0 | 99 | 99 | 50
Participants |  | 58 | 75 | 12
Statistical Analysis 1: Comparison: Sodium Zirconium Cyclosilicate (ZS) 5g vs Placebo; Treatment group comparisons were made using a logistic regression model containing the following covariates: treatment group; both baseline S-K values (48-hours open-label initial phase and double-blind randomized phase); baseline eGFR (during 48-hour open-label initial phase); age category (<55, 55-64, >=65 years); country; baseline RAAS inhibitor, chronic kidney disease, heart failure, and diabetes mellitus statuses; Test type: Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 6.3436, 95% CI 2-sided [2.6866 to 14.9782]
Statistical Analysis 2: Comparison: Sodium Zirconium Cyclosilicate (ZS) 10g vs Placebo; Test type: Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 18.1876, 95% CI 2-sided [7.1591 to 46.2054]

7. Secondary Outcome: Proportion of Normokalemic Patients at Day 1 Through Day 29/Exit
Description: The proportion of patients who are normokalemic (as defined by S-K between 3.5-5.0 mmol/l, inclusive) at Day 1 through Day 29/Exit in randomization phase. The results in the table below are presented for RTP.
Time Frame: Through 28-day randomized treatment phase.
Population: Full Analysis Set
Measure: Number; unit: Participants
Arm/Group | Sodium Zirconium Cyclosilicate (ZS) 10g Tid | Sodium Zirconium Cyclosilicate (ZS) 5g | Sodium Zirconium Cyclosilicate (ZS) 10g | Placebo
Number analyzed (Participants) | 0 | 99 | 99 | 50
Participants
  Day 1 |  | 93 | 94 | 45
  Day 2: number analyzed (Participants) | 0 | 98 | 98 | 50
  Day 2 |  | 89 | 93 | 40
  Day 5: number analyzed (Participants) | 0 | 98 | 98 | 50
  Day 5 |  | 71 | 89 | 27
  Day 8: number analyzed (Participants) | 0 | 95 | 98 | 49
  Day 8 |  | 62 | 81 | 16
  Day 12: number analyzed (Participants) | 0 | 93 | 96 | 48
  Day 12 |  | 62 | 78 | 12
  Day 15: number analyzed (Participants) | 0 | 92 | 93 | 48
  Day 15 |  | 57 | 77 | 12
  Day 19: number analyzed (Participants) | 0 | 90 | 91 | 46
  Day 19 |  | 55 | 76 | 11
  Day 22: number analyzed (Participants) | 0 | 87 | 90 | 43
  Day 22 |  | 54 | 73 | 11
  Day 26: number analyzed (Participants) | 0 | 88 | 91 | 42
  Day 26 |  | 56 | 74 | 8
  Day 29: number analyzed (Participants) | 0 | 86 | 88 | 41
  Day 29 |  | 51 | 71 | 11
  Day 29/Exit |  | 58 | 77 | 12

8. Secondary Outcome: Days Patients Remain Normokalemic
Description: The number of days patients remain normokalemic during the 28-day randomized treatment study phase. The results in the table below are presented for RTP.
Time Frame: Through 28-day randomized treatment phase.
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: Day
Arm/Group | Sodium Zirconium Cyclosilicate (ZS) 10g Tid | Sodium Zirconium Cyclosilicate (ZS) 5g | Sodium Zirconium Cyclosilicate (ZS) 10g | Placebo
Number analyzed (Participants) | 0 | 99 | 99 | 50
Day |  | 10.810 (1.113) | 15.623 (1.143) | 3.543 (1.351)
Statistical Analysis 1: Comparison: Sodium Zirconium Cyclosilicate (ZS) 5g vs Placebo; Results derived from a linear regression model with the following covariates: treatment group; baseline S-K values (Open-label phase and Randomized treatment phase); baseline eGFR; age category; country; baseline RAAS inhibitor, chronic kidney disease, heart failure, and diabetes mellitus statuses; Test type: Other; p < 0.001, Regression, Linear; Mean Difference (Final Values) = 7.266, 95% CI 2-sided [4.318 to 10.214]
Statistical Analysis 2: Comparison: Sodium Zirconium Cyclosilicate (ZS) 10g vs Placebo; Test type: Other; p < 0.001, Regression, Linear; Mean Difference (Final Values) = 12.079, 95% CI 2-sided [9.118 to 15.040]

9. Secondary Outcome: Mean Change in S-K Levels
Description: The mean change in S-K levels evaluated relative to both baselines. The results in the table below are presented for RTP.
Time Frame: Through 28-day randomized treatment phase.
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Sodium Zirconium Cyclosilicate (ZS) 10g Tid | Sodium Zirconium Cyclosilicate (ZS) 5g | Sodium Zirconium Cyclosilicate (ZS) 10g | Placebo
Number analyzed (Participants) | 0 | 99 | 99 | 50
mmol/L
  Day 2 change from RTP baseline: number analyzed (Participants) | 0 | 98 | 98 | 50
  Day 2 change from RTP baseline |  | 0.03 (0.354) | -0.09 (0.372) | 0.17 (0.443)
  Day 5 change from RTP baseline: number analyzed (Participants) | 0 | 98 | 98 | 50
  Day 5 change from RTP baseline |  | 0.23 (0.478) | -0.08 (0.439) | 0.60 (0.562)
  Day 8 change from RTP baseline: number analyzed (Participants) | 0 | 95 | 98 | 49
  Day 8 change from RTP baseline |  | 0.44 (0.487) | 0.00 (0.489) | 0.91 (0.622)
  Day 12 change from RTP baseline: number analyzed (Participants) | 0 | 93 | 96 | 48
  Day 12 change from RTP baseline |  | 0.53 (0.560) | 0.05 (0.573) | 0.97 (0.646)
  Day 15 change from RTP baseline: number analyzed (Participants) | 0 | 92 | 93 | 48
  Day 15 change from RTP baseline |  | 0.54 (0.584) | 0.04 (0.564) | 0.85 (0.585)
  Day 19 change from RTP baseline: number analyzed (Participants) | 0 | 90 | 91 | 46
  Day 19 change from RTP baseline |  | 0.56 (0.578) | 0.05 (0.576) | 0.97 (0.566)
  Day 22 change from RTP baseline: number analyzed (Participants) | 0 | 87 | 90 | 43
  Day 22 change from RTP baseline |  | 0.47 (0.555) | 0.10 (0.613) | 0.93 (0.702)
  Day 26 change from RTP baseline |  | 0.51 (0.581) | 0.05 (0.639) | 1.01 (0.607)
  Day 29 change from RTP baseline: number analyzed (Participants) | 0 | 86 | 88 | 41
  Day 29 change from RTP baseline |  | 0.47 (0.586) | 0.02 (0.665) | 1.02 (0.594)
  EOS change from RTP baseline: number analyzed (Participants) | 0 | 98 | 99 | 50
  EOS change from RTP baseline |  | 0.92 (0.661) | 0.77 (0.695) | 0.88 (0.684)
  Day 2 change from OLP baseline: number analyzed (Participants) | 0 | 98 | 98 | 50
  Day 2 change from OLP baseline |  | -1.28 (0.544) | -1.36 (0.515) | -1.07 (0.602)
  Day 5 change from OLP baseline: number analyzed (Participants) | 0 | 98 | 98 | 50
  Day 5 change from OLP baseline |  | -1.08 (0.552) | -1.35 (0.601) | -0.64 (0.594)
  Day 8 change from OLP baseline: number analyzed (Participants) | 0 | 95 | 98 | 49
  Day 8 change from OLP baseline |  | -0.87 (0.578) | -1.28 (0.634) | -0.34 (0.661)
  Day 12 change from OLP baseline: number analyzed (Participants) | 0 | 93 | 96 | 48
  Day 12 change from OLP baseline |  | -0.79 (0.603) | -1.21 (0.671) | -0.28 (0.602)
  Day 15 change from OLP baseline: number analyzed (Participants) | 0 | 92 | 93 | 48
  Day 15 change from OLP baseline |  | -0.77 (0.604) | -1.23 (0.643) | -0.40 (0.550)
  Day 19 change from OLP baseline: number analyzed (Participants) | 0 | 90 | 91 | 46
  Day 19 change from OLP baseline |  | -0.74 (0.639) | -1.20 (0.672) | -0.30 (0.533)
  Day 22 change from OLP baseline: number analyzed (Participants) | 0 | 87 | 90 | 43
  Day 22 change from OLP baseline |  | -0.84 (0.597) | -1.15 (0.730) | -0.38 (0.571)
  Day 26 change from OLP baseline: number analyzed (Participants) | 0 | 88 | 91 | 42
  Day 26 change from OLP baseline |  | -0.79 (0.687) | -1.21 (0.762) | -0.28 (0.563)
  Day 29 change from OLP baseline: number analyzed (Participants) | 0 | 86 | 88 | 41
  Day 29 change from OLP baseline |  | -0.82 (0.604) | -1.24 (0.734) | -0.27 (0.515)
  EOS change from OLP baseline: number analyzed (Participants) | 0 | 98 | 99 | 50
  EOS change from OLP baseline |  | -0.39 (0.649) | -0.50 (0.725) | -0.36 (0.702)

10. Secondary Outcome: Mean Percentage Change in S-K Levels
Description: The mean percentage change in S-K levels evaluated relative to both baselines. The results in the table below are presented for RTP.
Time Frame: Through 28-day randomized treatment phase.
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Sodium Zirconium Cyclosilicate (ZS) 10g Tid | Sodium Zirconium Cyclosilicate (ZS) 5g | Sodium Zirconium Cyclosilicate (ZS) 10g | Placebo
Number analyzed (Participants) | 0 | 99 | 99 | 50
Percentage change
  Day 2 percentage change from RTP baseline: number analyzed (Participants) | 0 | 98 | 98 | 50
  Day 2 percentage change from RTP baseline |  | 1.00 (8.459) | -1.74 (7.981) | 4.19 (10.592)
  Day 5 percentage change from RTP baseline: number analyzed (Participants) | 0 | 98 | 98 | 50
  Day 5 percentage change from RTP baseline |  | 5.51 (11.337) | -1.52 (9.691) | 14.19 (13.162)
  Day 8 percentage change from RTP baseline: number analyzed (Participants) | 0 | 95 | 98 | 49
  Day 8 percentage change from RTP baseline |  | 10.26 (11.340) | 0.16 (11.062) | 21.55 (15.634)
  Day 12 percentage change from RTP baseline: number analyzed (Participants) | 0 | 93 | 96 | 48
  Day 12 percentage change from RTP baseline |  | 12.41 (13.113) | 1.60 (13.205) | 22.87 (16.457)
  Day 15 percentage change from RTP baseline: number analyzed (Participants) | 0 | 92 | 93 | 48
  Day 15 percentage change from RTP baseline |  | 12.50 (13.378) | 1.27 (12.937) | 20.15 (14.647)
  Day 19 percentage change from RTP baseline: number analyzed (Participants) | 0 | 90 | 91 | 46
  Day 19 percentage change from RTP baseline |  | 13.12 (13.180) | 1.70 (13.139) | 22.77 (14.583)
  Day 22 percentage change from RTP baseline: number analyzed (Participants) | 0 | 87 | 90 | 43
  Day 22 percentage change from RTP baseline |  | 11.04 (12.993) | 2.66 (14.042) | 22.28 (18.131)
  Day 26 percentage change from RTP baseline |  | 12.02 (13.616) | 1.49 (14.441) | 23.63 (15.353)
  Day 29 percentage change from RTP baseline: number analyzed (Participants) | 0 | 86 | 88 | 41
  Day 29 percentage change from RTP baseline |  | 11.34 (13.821) | 0.87 (15.084) | 23.99 (15.329)
  EOS percentage change from RTP baseline: number analyzed (Participants) | 0 | 98 | 99 | 50
  EOS percentage change from RTP baseline |  | 21.62 (16.027) | 17.76 (16.266) | 20.70 (17.035)
  Day 2 percentage change from OLP baseline: number analyzed (Participants) | 0 | 98 | 98 | 50
  Day 2 percentage change from OLP baseline |  | -22.12 (8.679) | -23.55 (7.652) | -18.51 (9.751)
  Day 5 percentage change from OLP baseline: number analyzed (Participants) | 0 | 98 | 98 | 50
  Day 5 percentage change from OLP baseline |  | -18.77 (9.347) | -23.31 (9.230) | -10.96 (9.724)
  Day 8 percentage change from OLP baseline: number analyzed (Participants) | 0 | 95 | 98 | 49
  Day 8 percentage change from OLP baseline |  | -15.01 (9.627) | -22.01 (10.037) | -5.41 (11.424)
  Day 12 percentage change from OLP baseline: number analyzed (Participants) | 0 | 93 | 96 | 48
  Day 12 percentage change from OLP baseline |  | -13.55 (9.891) | -20.84 (10.981) | -4.57 (10.335)
  Day 15 percentage change from OLP baseline: number analyzed (Participants) | 0 | 92 | 93 | 48
  Day 15 percentage change from OLP baseline |  | -13.35 (10.170) | -21.18 (10.351) | -6.63 (9.457)
  Day 19 percentage change from OLP baseline: number analyzed (Participants) | 0 | 90 | 91 | 46
  Day 19 percentage change from OLP baseline |  | -12.79 (11.339) | -20.67 (10.834) | -4.89 (9.279)
  Day 22 percentage change from OLP baseline: number analyzed (Participants) | 0 | 87 | 90 | 43
  Day 22 percentage change from OLP baseline |  | -14.49 (10.158) | -19.67 (11.723) | -6.43 (9.759)
  Day 26 percentage change from OLP baseline: number analyzed (Participants) | 0 | 88 | 91 | 42
  Day 26 percentage change from OLP baseline |  | -13.35 (11.599) | -20.75 (12.360) | -4.74 (9.551)
  Day 29 percentage change from OLP baseline: number analyzed (Participants) | 0 | 86 | 88 | 41
  Day 29 percentage change from OLP baseline |  | -14.09 (9.949) | -21.42 (11.659) | -4.61 (8.802)
  EOS percentage change from OLP baseline: number analyzed (Participants) | 0 | 98 | 99 | 50
  EOS percentage change from OLP baseline |  | -6.57 (11.199) | -8.54 (12.405) | -5.95 (11.927)

11. Secondary Outcome: Number of Hyperkalemic Patients
Description: The results represent number of hyperkalemic patients during the 28-day randomized treatment study phase. The results in the table below are presented for RTP.
Time Frame: Through 28-day randomized treatment phase.
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Sodium Zirconium Cyclosilicate (ZS) 10g Tid | Sodium Zirconium Cyclosilicate (ZS) 5g | Sodium Zirconium Cyclosilicate (ZS) 10g | Placebo
Number analyzed (Participants) | 0 | 99 | 99 | 50
Participants |  | 66 | 45 | 47
Statistical Analysis 1: Comparison: Sodium Zirconium Cyclosilicate (ZS) 5g vs Placebo; Results derived from a Cox Proportional Hazards model with the following covariates: treatment group, both baseline S-K values (48-hours open-label initial phase and double-blind randomized phase), baseline eGFR, age category (<55, 55-64, >=65 years), country, baseline RAAS inhibitor, chronic kidney, disease heart failure, and diabetes mellitus statuses; Test type: Other; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 0.443, 95% CI 2-sided [0.2954 to 0.6631]
Statistical Analysis 2: Comparison: Sodium Zirconium Cyclosilicate (ZS) 10g vs Placebo; Test type: Other; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 0.158, 95% CI 2-sided [0.0992 to 0.2508]

12. Secondary Outcome: Mean Changes in S-Aldosterone and P Renin Levels
Description: The mean changes from OLP baseline in S-Aldosterone and P-Renin levels. The results in the table below are presented for RTP.
Time Frame: Through 28-day randomized treatment phase.
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Sodium Zirconium Cyclosilicate (ZS) 10g Tid | Sodium Zirconium Cyclosilicate (ZS) 5g | Sodium Zirconium Cyclosilicate (ZS) 10g | Placebo
Number analyzed (Participants) | 0 | 99 | 99 | 50
pmol/L
  Day 1 S-Aldosterone: number analyzed (Participants) | 0 | 89 | 83 | 46
  Day 1 S-Aldosterone |  | -112.69 (178.358) | -85.63 (118.017) | -98.54 (168.657)
  Day 15 S-Aldosterone: number analyzed (Participants) | 0 | 82 | 77 | 46
  Day 15 S-Aldosterone |  | -91.75 (179.791) | -96.37 (108.002) | 39.78 (152.050)
  Day 29 S-Aldosterone: number analyzed (Participants) | 0 | 76 | 68 | 40
  Day 29 S-Aldosterone |  | -102.70 (212.187) | -90.22 (91.149) | 41.07 (198.266)
  Day 1 P-Renin: number analyzed (Participants) | 0 | 91 | 92 | 47
  Day 1 P-Renin |  | -0.23 (1.158) | -0.26 (1.913) | -0.30 (1.031)
  Day 15 P-Renin: number analyzed (Participants) | 0 | 80 | 81 | 44
  Day 15 P-Renin |  | -0.39 (1.350) | -1.09 (4.732) | 0.60 (3.250)
  Day 29 P-Renin: number analyzed (Participants) | 0 | 75 | 78 | 37
  Day 29 P-Renin |  | -0.27 (1.008) | -1.56 (4.165) | -0.25 (2.725)

13. Secondary Outcome: Patient Reported Health State (EQ-5D) Questionnaire
Description: Evaluate health state of patients using EQ-5D questionnaire. This scale is numbered from 0 to 100. 0 means the worst health you can imagine. 100 means the best health you can imagine. The results in the table below are presented for RTP.
Time Frame: Through study completion, an average of 37 days.
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Sodium Zirconium Cyclosilicate (ZS) 10g Tid | Sodium Zirconium Cyclosilicate (ZS) 5g | Sodium Zirconium Cyclosilicate (ZS) 10g | Placebo
Number analyzed (Participants) | 0 | 99 | 99 | 50
Units on a scale
  OLP baseline: number analyzed (Participants) | 0 | 91 | 88 | 43
  OLP baseline |  | 75.0 (16.44) | 74.3 (17.44) | 72.7 (17.32)
  Day 29: number analyzed (Participants) | 0 | 86 | 88 | 41
  Day 29 |  | 77.6 (16.50) | 76.9 (16.08) | 76.6 (14.08)

ADVERSE EVENTS:
Time Frame: Through 28-day randomized treatment study phase day 8-29
Arm/Group | Sodium Zirconium Cyclosilicate (ZS) 10g Tid | Sodium Zirconium Cyclosilicate (ZS) 5g | Sodium Zirconium Cyclosilicate (ZS) 10g | Placebo
All-Cause Mortality (participants affected / at risk) | 0/267 | 0/99 | 0/99 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/267 | 4/99 | 3/99 | 1/50
Other Adverse Events (participants affected / at risk) | 0/267 | 6/99 | 21/99 | 0/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sodium Zirconium Cyclosilicate (ZS) 10g Tid (N=267) | Sodium Zirconium Cyclosilicate (ZS) 5g (N=99) | Sodium Zirconium Cyclosilicate (ZS) 10g (N=99) | Placebo (N=50)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infectious colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sodium Zirconium Cyclosilicate (ZS) 10g Tid (N=267) | Sodium Zirconium Cyclosilicate (ZS) 5g (N=99) | Sodium Zirconium Cyclosilicate (ZS) 10g (N=99) | Placebo (N=50)
Oedema peripheral (General disorders) | 0 (0) | 4 (4) | 7 (7) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 9 (9) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1) | 8 (9) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-03-15): https://cdn.clinicaltrials.gov/large-docs/34/NCT02875834/SAP_000.pdf
  • Study Protocol (2017-09-22): https://cdn.clinicaltrials.gov/large-docs/34/NCT02875834/Prot_001.pdf